CLINICAL TRIAL: NCT04800991
Title: A Pilot Study to Evaluate the Feasibility and Efficacy of Digital Health Technology for Postoperative Care With Gastrectomy-Treated Patients in Gastric Cancer
Brief Title: NuGa (Nutrition for Gastric Cancer Patients)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Kwang Yang, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HDT-202_F01
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Gastric Cancer
Keywords: Gastrectomy; postoperative care; nutrition; Digital health technology; Application
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: HDT-202(application)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhexium Onco Nutrition(HDT-202) (Experimental): "subject mobile application" and "Investigator web portal" with no invasive action on the human body
  Interventions: Device: Rhexium Onco Nutrition

INTERVENTIONS:
Device: Rhexium Onco Nutrition — The research devices in this study are classified into "subject mobile application" and "investigator web portal" with no invasive action on the human body
  Other Names: HDT-202

SUMMARY:
The objective of this pilot study is to evaluate the feasibility and efficacy of Rhexium Onco Nutrition, HDT-202 for post-operative care in patients who have undergone gastrectomy.

DETAILED DESCRIPTION:
1. A total of 4 visits will be performed.
2. At the screening visit,subject's written informed consent, assessing the inclusion/exclusion criteria and assigning enrollment numbers to eligible subjects, demographic information taking, medical history/medication history taking, vital signs measuring, physical examination, height and body weight measuring, instructing how to install/use the investigational device, and administering quality of life questionnaires.
3. During the treatment period, a total of 3 visits will be performed. To evaluate feasibility and efficacy, the following procedures will be carried out: vital signs measuring, physical examination, nutrition assessment/consultation, evaluation of feasibility for 'subjects', evaluation of feasibility for 'investigators', and adverse events (AEs)/concomitant medications checking and collecting.
4. During the treatment period, telephone monitoring is conducted depending on the compliance of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who voluntarily signs the informed consent form for this study
2. Age of ≥19 years old
3. Patient who has undergone therapeutic gastrectomy after a diagnosis of gastric cancer
4. Able to eat food orally after gastrectomy
5. Patient who possesses an Android OS based mobile device and is capable of using the investigational device.

Exclusion Criteria:

1. Other cancer or metastasis documented within 5 years prior to screening
2. Ongoing or planned enteral tube feeding or total parenteral nutrition
3. Other clinically significant medical or psychiatric findings based on which the individual is considered by the investigator to be ineligible
4. Individual who possesses a mobile device on which the application is unable to be installed and/or run normally for technical reasons
5. Individual who, in the opinion of the investigator, has difficulty understanding how to use the investigational device or is unlikely to comply with other study procedures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Score of each domain of the 'feasibility assessment of the investigational device (application)' questionnaire for subjects | Week 2 (Visit 2)
  higher scores mean a better outcome
Score of each domain of the 'feasibility assessment of the investigational device (application)' questionnaire for subjects | Week 6 (Visit 3),
  higher scores mean a better outcome
Score of each domain of the 'feasibility assessment of the investigational device (application)' questionnaire for subjects | Week 10 (Visit 4)
  higher scores mean a better outcome
Score of each domain of the 'feasibility assessment of the investigational device (website)' questionnaire for investigators | Week 6 (Visit 3)
  higher scores mean a better outcome

SECONDARY OUTCOMES:
Change from baseline (Visit 1) in 'EORTC QLQ-C30' score | baseline (Visit 1), Week 10 (Visit 4)
  Refer to Title
Change from baseline (Visit 1) in 'EORTC QLQ-STO22' score | baseline (Visit 1), Week 10 (Visit 4)
  Refer to Title
Change from baseline (Visit 1) in 'KOQUSS Index' score | baseline (Visit 1), Week 10 (Visit 4)
  Refer to Title
Correlation between change from Day 1 in body weight at Week 10 (Visit 4) and calory goal achievement rate | Week 10 (Visit 4)
  Refer to Title
Correlation between change from Day 1 in body weight at Week 10 (Visit 4) and protein intake goal achievement rate | Week 10 (Visit 4)
  Refer to Title
Frequency of each symptom between visits after using the investigational device (application) | Week 2 (Visit 2), Week 6 (Visit 3), Week 10 (Visit 4)
  Refer to Title
The investigational device(application) usage compliance by age | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by gender | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by surgery | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by stage of disease | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by body mass index [BMI] before discharge from hospital | Week 10 (Visit 4)
  weight and height will be combined to report BMI in kg/m^2, compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by status of postoperative anticancer therapy | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100
The investigational device(application) usage compliance by underlying disease | Week 10 (Visit 4)
  compliance(%) will be measured to day of usage/total period*100

OTHER OUTCOMES:
Frequency of each symptom by baseline characteristics (age, gender, surgery, stage of disease, BMI before discharge from hospital, status of postoperative anticancer therapy, underlying disease) | Week 10 (Visit 4)
  Refer to Title
Frequency of Adverse Events | Week 2 (Visit 2), Week 6 (Visit 3), Week 10 (Visit 4)
  Incident rate of Adverse Events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Han-Kwang Yang, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Surgery, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JH, Lee HJ, Kim J, Cho YS, Lee S, Park S, Choe H, Song E, Kim Y, Kong SH, Park DJ, Nam BH, Yang HK. Development and Feasibility Assessment of Mobile Application-Based Digital Therapeutics for Postoperative Supportive Care in Gastric Cancer Patients Following Gastrectomy. J Gastric Cancer. 2024 Oct;24(4):420-435. doi: 10.5230/jgc.2024.24.e37. PMID 39375057